CLINICAL TRIAL: NCT00751517
Title: Cyclophosphamide Versus Methotrexate for Remission Maintenance in Systemic Necrotizing Vasculitides. A Randomized Controlled Trial.
Brief Title: Cyclophosphamide Versus Methotrexate for Remission Maintenance in Systemic Necrotizing Vasculitides
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Parma (Other)
Responsible Party: Carlo Buzio, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCM 01
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Wegener's Granulomatosis; Churg-Strauss Syndrome; Microscopic Polyangiitis; Polyarteritis Nodosa
Keywords: Vasculitis; Cyclophosphamide; Methotrexate; Systemic Necrotizing Vasculitides
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Churg-Strauss Syndrome; Microscopic Polyangiitis; Polyarteritis Nodosa; Vasculitis | interventions — Methotrexate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Cyclophosphamide
  Interventions: Drug: Cyclophosphamide
- B (Experimental): Methotrexate
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate
  Arms: B
Drug: Cyclophosphamide
  Arms: A

SUMMARY:
The Systemic Necrotizing Vasculitides (SNV) encompass a group of rare diseases which include Wegener's Granulomatosis (WG), Churg-Strauss Syndrome (CSS), Microscopic polyangiitis (MPA)and Polyarteritis nodosa (PAN). Common histological findings are inflammation with fibrinoid necrosis of the small vessels and sporadic or absent immune-deposits. The gold standard therapy for SNV is currently represented by the association of Cyclophosphamide and Prednisone. The limits of this approach are the high frequency of recurrent disease and an increased incidence of malignancy and infections. The aim of the present study is to compare the efficacy of Methotrexate vs Cyclophosphamide for Remission Maintenance in SNV.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically active SNV
* Life-expectancy > 1 year
* Written informed consent

Exclusion Criteria:

* Creatinine clearance < 10 ml/min/1.73 mq
* Aminotransferase levels more than twice the upper limit of the normal range
* HBsAg positivity
* anti-HCV Ig and HCV-RNA positivity
* HIV positivity
* Active malignancies
* Coexistence of connective tissue disease
* Prednisolone, cyclophosphamide or methotrexate hypersensitivity
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Time from remission to relapse

SECONDARY OUTCOMES:
Recurrence rate
Therapy-related toxicity
Hospitalization rate
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Buzio, MD, Principal Investigator — University of Parma
Locations (1):
- Department of Clinical Medicine Nephrology and Health Science, Parma University Hospital, Parma, Italy/Parma, Italy

REFERENCES:
- [Background] Hoffman GS, Kerr GS, Leavitt RY, Hallahan CW, Lebovics RS, Travis WD, Rottem M, Fauci AS. Wegener granulomatosis: an analysis of 158 patients. Ann Intern Med. 1992 Mar 15;116(6):488-98. doi: 10.7326/0003-4819-116-6-488. PMID 1739240
- [Background] Hoffman GS. Wegener's granulomatosis. Curr Opin Rheumatol. 1993 Jan;5(1):11-7. doi: 10.1097/00002281-199305010-00003. PMID 8435284
- [Background] Gordon M, Luqmani RA, Adu D, Greaves I, Richards N, Michael J, Emery P, Howie AJ, Bacon PA. Relapses in patients with a systemic vasculitis. Q J Med. 1993 Dec;86(12):779-89. PMID 7906421
- [Background] Falk RJ, Jennette JC. ANCA small-vessel vasculitis. J Am Soc Nephrol. 1997 Feb;8(2):314-22. doi: 10.1681/ASN.V82314. No abstract available. PMID 9048352
- [Background] Talar-Williams C, Hijazi YM, Walther MM, Linehan WM, Hallahan CW, Lubensky I, Kerr GS, Hoffman GS, Fauci AS, Sneller MC. Cyclophosphamide-induced cystitis and bladder cancer in patients with Wegener granulomatosis. Ann Intern Med. 1996 Mar 1;124(5):477-84. doi: 10.7326/0003-4819-124-5-199603010-00003. PMID 8602705
- [Derived] Maritati F, Alberici F, Oliva E, Urban ML, Palmisano A, Santarsia F, Andrulli S, Pavone L, Pesci A, Grasselli C, Santi R, Tumiati B, Manenti L, Buzio C, Vaglio A. Methotrexate versus cyclophosphamide for remission maintenance in ANCA-associated vasculitis: A randomised trial. PLoS One. 2017 Oct 10;12(10):e0185880. doi: 10.1371/journal.pone.0185880. eCollection 2017. PMID 29016646